CLINICAL TRIAL: NCT05585294
Title: The Effectiveness of Perturbation Exercises in Elderly Back Pain
Brief Title: Water Versus Land Based Perturbation Exercises in Elderly Participants With Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gulf Medical University (Other)
Collaborators: Srinivas University (Unknown)
Responsible Party: Principal Investigator, Rania Zaarour, Assistant Professor, Gulf Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: INT/COHS/UG/012-2019; COHS_UG_Research_6122017 (Other: GMU Ethical commitee)
Record Dates: First submitted 2022-10-13; First posted 2022-10-18 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Back Pain; Back Pain With Radiation; Back Pain Without Radiation; Back Pain Lower Back Chronic
Keywords: Back Pain; Old Age; Exercises; Hydrotherapy; Rehabilitation
MeSH Terms: conditions — Back Pain; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: pre and post outcomes comparison after clinical intervention
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Outcome assessor unaware of what care was provided, and care was provided by other providers. Possibility of sequential trail is considered. The value of p will be adjusted depending the number of analysis made and stopping rule will be followed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Water based perturbation exercise group (Experimental): In both groups, the participants screened for Treatment-based classification of back pain and based on TBC interventions were provided. From second week, water based perturbation exercise were initiated personalized to the level of participants.
  Treatment-based classification of back pain intervention was gradually tapered in orderly fashion during 6 weeks, concurrently introduced land based perturbation exercise gradually phased from level 1 to level 4.
  Interventions: Behavioral: Exercises
- Land based perturbation exercise group (Active Comparator): All procedures were followed similar to Water based perturbation exercise group except perturbation based exercises were provided in land.
  Interventions: Behavioral: Exercises

INTERVENTIONS:
Behavioral: Exercises — Perturbation exercises: A new protocol of perturbation exercises aimed to disturb static and dynamic posture or equilibrium at primarily at body segments at hip and shoulder level were provided. The perturbation was initially started as anticipatory postural adjustment and progressed to compensatory postural adjustment, where stepping on various directions were challenged. The nature of perturbation or push or nudges applied by physiotherapists were progressed from a) self-generated to therapist applied, anticipated to unanticipated, stable to unstable platforms, static to dynamic postural tasks with loaded extremities and at higher level simple to higher cognitive tasks were also incorporated.
  Other Names: Mckenzie extension exercise, mobilization and spinal lumbar traction therapy tailored based on TBC system

SUMMARY:
The aim of this study was to compare the effectiveness of land based versus water based perturbation exercises on the pain, disability, fear of falling, and fear avoidance beliefs in elderly participants. Overweight/obese subgroup was compared with healthy weight with chronic low back pain participants to investigate any effect on BMI on both interventions. The results of the study revealed that both exercise groups i.e., land and water based exercise had a significant reduction in pain level, fear of falling, fear avoidance belief related to work, disability and improved SLR.

DETAILED DESCRIPTION:
Twenty-four grouped into 12 per group participated water based and land based exercise protocol. Both groups were given McKenzie Method of exercises in 1st week based on the treatment-based classification (TBC) approach or personalized to the need of participants as per TBC.

Perturbation-based postural exercises were given to participants, which were performed on land or water for 6 weeks.

The perturbation based exercises were categorized into four levels, where level 1:static postural control, 2:dynamic postural control 3:Extremity loaded postural control and 4: cognitive task associated postural control. The perturbation were provided at shoulder and hip level, by intervention providers progressive enough to initiate anticipatory or compensatory postural adjustments.

Both groups were educated on pain assurance and spinal ergonomics feedback. The Outcomes were measured using a Visual analog scale, Oswestry disability index, Fear avoidance belief questionnaire, Straight leg raise, Modified fall efficacy scale, and Borg scale. The pain level were assessed for personalized progression from level 1 to level 4 progression of perturbation exercises.

Both the exercise groups of land and water showed improvement in measured clinical outcomes in terms of reduction in pain level, fear of falling, fear avoidance belief related to work, SLR, and disability. Water-based group showed additional benefits and significant improvement in fear avoidance belief related to physical activity and exercised with low rate of perceived exertion.

ELIGIBILITY:
Inclusion Criteria:

* Pain history of minimum 12 weeks duration in below labels
* Participants with the diagnostic labels of spondylosis
* Non-specific chronic low back pain
* Back pain radiating to leg or sciatica
* Subacute back pain

Exclusion Criteria:

* Unstable blood pressure
* Cardiac failure
* Incontinence
* Uncontrolled epilepsy
* Open wounds
* Acute infections
* Neurological disorders
* Orthopedic conditions affecting exercise participation in pool and land
* Cardio-respiratory conditions affecting exercise participation in pool and land.

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-12-21 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Low back pain | 6 weeks
  Visual Analogue Scale (VAS) was used where 0 indicates no pain and 10 indicate extremely painful.
Disability caused by the chronic low back pain | 6 weeks
  A standard Oswestry Disability Index (ODI) was used to evaluate the disability caused by the chronic low back pain. The lower the score lower disability and higher scores indicates that high level of disability associated with back pain.
Physical activity associated fear avoidance behavior | 6 weeks
  The percentage of fear avoidance of behavior ranges from 0 to 100% where 0%-indicates no fear and 100%-indicate highest level of fear avoidance behavior.
Fall risk | 6 weeks
  Fall risk of participants was assessed using the Modified fall efficacy scale (MFES), where Higher scores reflect more confidence and less fear of falling while lower scores reflect less confidence and more fear of falling.

SECONDARY OUTCOMES:
Rate of perceived exertion | 6 weeks
  Borg scale utilised to measue the exertion during the exercise. Grades were obtained with 6 being no exertion at all, and 20 being maximum effort.
Impairment - Straight Leg Raise as hip joint range of motion | 6 weeks
  Straight leg raise range of motion was measured to identify the level of impairment and to confirm any leg pain associated with back pain

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Ramprasad Muthukrishnan, Ph.D, Principal Investigator — Gulf Medical Univesity
Locations (2):
- United Arab Emirates (2):
  - Gulf Medical University, Thumbay Physical Therapy and Rehabiliation Hospital, Thumbay University Hospital, Ajman
  - Gulf Medical University, Ajman

IPD SHARING:
Plan to Share IPD: Yes
Upon receipt of a request from other parties, for scientific purposes such as Systematic review and meta-analysis, the data will be shared, without disclosing the personal data.
Supporting Information: Study Protocol, CSR
Time Frame: The data is available and processed final.
Access Criteria: Upon receipt of a request from other parties, for scientific purposes such as Systematic review and meta-analysis, the data will be shared, without disclosing the personal data.

REFERENCES:
- [Derived] Muthukrishan R, Badr Ul Islam FM, Shanmugam S, Arulsingh W, Gopal K, Kandakurti PK, Rajasekar S, Malik GS, S G G. Perturbation-based Balance Training in Adults Aged Above 55 Years with Chronic Low Back Pain: A Comparison of Effects of Water versus Land Medium - A Preliminary Randomized Trial. Curr Aging Sci. 2024;17(2):156-168. doi: 10.2174/0118746098254991231125143735. PMID 38111118